CLINICAL TRIAL: NCT02884661
Title: Assessment of the Usual Choice for a First-line Treatment in Case of Atrial Fibrillation : Comparison Between Cardiology Department and Geriatric Unit.
Brief Title: First-line Treatment for Atrial Fibrillation in Cardiology and Geriatric Departments
Acronym: ACFA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-05Obs-CHRMT
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hospitalization in Cardiology department: Patients cared by the Cardiology department
- Hospitalization in Geriatric unit: Patients cared by the Geriatric unit

SUMMARY:
In order to evaluate the implementation for the recommendations about the patient care for atrial fibrillation in aged patients, a non-interventional study is performed retrospectively by comparing two approach of the focus in Cardiology Department and in Geriatric unit.

ELIGIBILITY:
Inclusion Criteria:

* having an atrial fibrillation
* cared in Cardiology department or in geriatric unit

Exclusion Criteria:

* having a mitral valvulopathy, or a valvular disease with a surgery indication
* having a valvular prosthesis
* history of valve reconstruction

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with an atrial fibrillation and hospitalized in Cardiology department or in geriatric unit
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Implementation of the recommendations about non-valvular atrial fibrillation | September 1st, 2014 to October 13, 2015

SECONDARY OUTCOMES:
Socio-demographic data | September 1st, 2014 to October 13, 2015
Etiologic factors of the atrial fibrillations | September 1st, 2014 to October 13, 2015
Use of supplementary examinations | September 1st, 2014 to October 13, 2015
Use of a standard geriatric assessment | September 1st, 2014 to October 13, 2015
Use of an assessment of the risks of thrombosis and bleeding | September 1st, 2014 to October 13, 2015
Choice of the anti-thrombosis treatment | September 1st, 2014 to October 13, 2015
Choice of the anti-arrhythmia treatment | September 1st, 2014 to October 13, 2015

CONTACTS AND LOCATIONS:
Overall Officials: NOEL BLETTNER, MD, Principal Investigator — CHR Metz-Thionville
Locations (1):
- CHR Metz-Thionville, Metz, France